CLINICAL TRIAL: NCT05540808
Title: Diagnostic Test of Full-targeted Pathogen Capture Metagenomics Next Generation Sequencing in Etiological Diagnosis of Sepsis
Brief Title: The Value of Full-targeted Pathogen Capture Metagenomics Next Generation Sequencing in Etiological Diagnosis of Sepsis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shenzhen Second People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20223357008
Record Dates: First submitted 2022-09-13; First posted 2022-09-15 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2022-07

CONDITIONS: Sepsis, Severe
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The etiological diagnosis of sepsis is the key to guide clinical treatment. Metagenomic sequencing (mNGS) is very suitable for the diagnosis of sepsis due to its rapid, accurate and not easy to be disturbed by the environment. However, the conventional pathogen mNGS has potential risks such as low detection rate, loss of intracellular bacteria and fungi. At present, the latest fully targeted pathogen capture mNGS technology makes up for the shortcomings of conventional methods by bidirectional enrichment of pathogen nucleic acids. The aim of this study was to explore the value of fully targeted pathogen capture mNGS in improving etiological diagnosis in patients with sepsis compared with conventional methods.

DETAILED DESCRIPTION:
This study planned to continuously collect samples from patients with sepsis who were admitted to the intensive care Unit of our hospital from 2022.08 to 2024.07, and conduct whole-target pathogen capture mNGS detection and follow-up etiological diagnosis based on blind method. The clinical diagnosis with clear etiology was taken as the gold standard.

ELIGIBILITY:
Inclusion Criteria:

* Critical care patients aged ≥ 18 years old
* Patients with sepsis

Exclusion Criteria:

* Lack of traditional pathogen detection results
* Discharge diagnosis without clear etiology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with sepsis
Sampling Method: Probability Sample
Enrollment: 86 (Estimated)
Dates: Start 2023-02-10 (Estimated); Primary Completion 2024-07-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
sensitivity | up to 3 year
  The chance of testing positive for a pathogen in a sample judged by the gold standard
specificity | up to 3 year
  The chance of a negative test in a sample judged pathogen-free by the gold standard

CONTACTS AND LOCATIONS:
Overall Officials: Ying Li, Study Chair — Shenzhen Second People's Hospital

IPD SHARING:
Plan to Share IPD: No